CLINICAL TRIAL: NCT05300165
Title: Role of Gut Microbiome in the Health Benefits
Acronym: BEEROTA18
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BEEROTA18
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Normal Population
Keywords: beer
MeSH Terms: interventions — Beer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal population (Other): 20 participants representing a normal population will include a daily beer in their meals, changing the kind of beer every 2 weeks from alcohol-free lager beer, lager beer, or dark beer.
  Interventions: Dietary Supplement: Beer

INTERVENTIONS:
Dietary Supplement: Beer — A daily beer will be consumed by the participants during a total of 6 weeks, changing every 2 weeks from alcohol-free lager beer, lager beer and dark beer

SUMMARY:
Beneficial effects of moderate chronic consumption of beer have been extensively reported, however, the mechanisms have not been elucidated yet. Gut microbiota is an important mediator in the homeostasis of the host. Polyphenols act as bacterial substrates and modulators of the gut microbiota. Indeed, the investigators have previously observed that the chronic moderate consumption of red wine by metabolic syndrome patients triggered in an amelioration of the metabolic syndrome variables, and this effect was mediated, at least partially, by the interaction of the gut microbiota with the polyphenols of the red wine. In this manner, beer has a medium content of polyphenols. Thus, the investigators propose that the beneficial effects of moderate chronic consumption of beer could be because of the action of the gut microbiota with the beer polyphenols. The investigators are going to perform an intervention study in which normal volunteers will consume three different beer types with different content in polyphenols and it will be analyzed the gut microbiota profile (Metagenomics), metabolites (Metabolomics) and metabolic syndrome markers (gene expression, ELISA) to establish the correspondent relationships, trying to decipher the implication of the gut microbiota in the beneficial effects of moderate chronic consumption of beer.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Usual consumer of Beer

Exclusion Criteria:

* being a non usual beer-consumer,
* body mass index (BMI) > 40 kg m2.
* acute or chronic infection, inflammatory disease or endocrine disorders; history of cancer; leukocytosis; anti-inflammatory, corticosteroid or hormone treatment.
* history of alcohol abuse or drug dependence.
* under a restrictive diet or a weight change ≥5 kg during the 3 months prior to the study.
* antibiotic therapy, prebiotics, probiotics, synbiotics, vitamin supplements or any other medical treatment influencing intestinal microbiota during the 3 months before the start of the study or during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota | Baseline, 2nd, 4th and 6th weeks visits
  change from baseline in 16S rRNA amplicons determined in DNA from feces after 6 weeks

SECONDARY OUTCOMES:
Change in caloric consumption | Baseline and 6th weeks visits
  change from baseline in the number of caloric consumption measured by an structured nutrient intake
Change in waist circumference | Baseline and 6th weeks visits
  Change from baseline in waist circumference (cm) after the completion of the trial
Change in glucose concentration | Baseline and 6th weeks visits
  Change from baseline in serum glucose level after the completion of the trial
Change in HDL-cholesterol concentration | Baseline and 6th weeks visits
  Change from baseline in serum HDL-cholesterol level after the completion of the trial
Change in triglycerides concentration | Baseline and 6th weeks visits
  Change from baseline in serum triglycerides level after the completion of the trial
Change in blood pressure | Baseline and 6th weeks visits
  Change from baseline in blood pressure (systolic and diastolic) after the completion of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J. Tinahones, PhD, Principal Investigator — Instituto de Investigacion Biomedica de Malaga
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Spain